CLINICAL TRIAL: NCT00045227
Title: A Pilot Trial of Pox Vector PSA Vaccine With Concurrent Docetaxel Versus Pox Vector Vaccine Followed by Docetaxel in Metastatic Androgen Independent Prostate Cancer
Brief Title: Vaccine Therapy With or Without Docetaxel in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000256919; NCI-02-C-0218; NCI-5319; NCT00041522 (obsolete NCT alias)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2003-12

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PROSTVAC; sargramostim; Docetaxel

INTERVENTIONS:
Biological: recombinant fowlpox-prostate specific antigen vaccine
Biological: recombinant vaccinia prostate-specific antigen vaccine
Biological: recombinant vaccinia-B7.1 vaccine
Biological: sargramostim
Drug: docetaxel

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining vaccine therapy with chemotherapy may kill more tumor cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of vaccine therapy with or without docetaxel in treating patients who have metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the relative change in prostate-specific antigen (PSA)-specific T-cell precursors (CD8) from baseline to day 85 in patients with metastatic androgen-independent prostate cancer treated with a vaccination regimen comprising fowlpox-PSA vaccine, recombinant rV-B7.1 vaccine, recombinant vaccinia-PSA vaccine, and sargramostim (GM-CSF) with or without docetaxel.
* Compare the safety of these regimens in these patients.
* Compare clinical activity of these regimens in these patients.
* Determine the immunologic effects in these patients after additional vaccine/chemotherapy courses.
* Measure CD4 T-cell responses to the vaccine in these patients.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms after receiving priming vaccinations.

* Priming vaccinations: All patients receive recombinant vaccinia-prostate-specific antigen (PSA) vaccine subcutaneously (SC) and recombinant rV-B7.1 vaccine SC on day 1 and sargramostim (GM-CSF) SC on days 1-4. Patients then receive fowlpox-PSA vaccine (F-PSA) SC on day 15 and GM-CSF SC on days 15-18.
* Arm I: Patients receive docetaxel IV over 30 minutes on days 29, 36, and 43; F-PSA SC on day 30; and GM-CSF SC on days 30-33. Treatment repeats beginning on day 56 for one more course. Patients who do not have disease progression at day 85 receive docetaxel weekly for 3 weeks and F-PSA on day 1 of each course. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive F-PSA SC on days 29 and 57 and GM-CSF SC on days 29-32 and 57-60. Patients who show disease progression after day 85 either radiographically or by rising PSA stop receiving the vaccine and may receive docetaxel weekly for 3 weeks. Chemotherapy repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 28 patients (14 per treatment arm) will be accrued for this study within 9-10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of androgen-independent metastatic adenocarcinoma of the prostate, confirmed by 1 of the following:

  * Histologically confirmed disease
  * Pathologically documented disease and clinical course consistent with prostate cancer
* Castrate levels of testosterone with progressive disease by at least 1 of the following parameters:

  * 2 consecutively rising prostate-specific antigen levels, separated by at least 1 week, with at least 1 measurement that is 50% above the nadir reached after the last therapeutic maneuver (must be at least 5 ng/mL)
  * At least 1 new metastatic deposit on technetium Tc 99 bone scintigraphy
  * Progression of soft-tissue metastases by imaging or palpation, as indicated by:

    * Development of new area of malignant disease
    * At least 20% increase in sum of the longest dimension of target lesions
* Serum testosterone less than 50 ng/dL if no prior surgical castration

  * Luteinizing hormone-releasing hormone therapy must continue
* HLA-A2 positive
* No brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 6 months

Hematopoietic

* Granulocyte count at least 1,500/mm^3
* Lymphocyte count at least 500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin less than 1.5 mg/dL
* AST and ALT less than 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN OR
* Hepatic alkaline phosphatase fraction less than 2.5 times ULN

Renal

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 40 mL/min
* Proteinuria grade 0-1 OR
* Protein less than 1,000 mg by 24-hour urine collection
* No hematuria
* No abnormal sediment unless non-renal

Cardiovascular

* No unstable or newly diagnosed angina pectoris
* No myocardial infarction within the past 6 months
* No New York Heart Association class II-IV congestive heart failure
* No concurrent clinically significant cardiomyopathy requiring treatment

Immunologic

* No prior allergy or untoward reaction to vaccinia virus vaccination
* No altered immune function, including:

  * Eczema
  * Atopic dermatitis
  * HIV
  * Autoimmune disease

    * Autoimmune neutropenia
    * Thrombocytopenia
    * Hemolytic anemia
    * Systemic lupus erythematosus
    * Sjogren's syndrome
    * Scleroderma
    * Myasthenia gravis
    * Goodpasture syndrome
    * Addison's disease
    * Hashimoto's thyroiditis
    * Active Graves' disease
    * Multiple sclerosis
* No extensive psoriasis, severe acneiform rash, impetigo, varicella zoster, burns, or other traumatic or pruritic skin condition
* No known allergy to eggs

Other

* No other malignancy within the past 2 years except nonmelanoma skin cancer or carcinoma in situ of the bladder
* No other life-threatening or serious illness
* No unhealed surgical scars
* No household or close physical contact with persons with any of the following conditions during or for 2 weeks after study treatment:

  * Eczema or eczematoid skin disorders
  * Acute, chronic, or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds)
  * Pregnant or nursing women
  * Children under 5 years of age
  * Immunodeficient or immunosuppressed (including HIV positive) individuals
* No history of seizures or encephalitis

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior taxanes for metastatic prostate cancer

Endocrine therapy

* See Disease Characteristics
* At least 4 weeks since prior flutamide
* At least 6 weeks since prior bicalutamide or nilutamide
* No concurrent steroids except topical steroids, inhaled steroids for mild or moderate asthma, or decadron as premedication for chemotherapy

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics
* No prior splenectomy

Other

* Recovered from prior therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-08; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip M. Arlen, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Result] Arlen PM, Gulley JL, Parker C, Skarupa L, Pazdur M, Panicali D, Beetham P, Tsang KY, Grosenbach DW, Feldman J, Steinberg SM, Jones E, Chen C, Marte J, Schlom J, Dahut W. A randomized phase II study of concurrent docetaxel plus vaccine versus vaccine alone in metastatic androgen-independent prostate cancer. Clin Cancer Res. 2006 Feb 15;12(4):1260-9. doi: 10.1158/1078-0432.CCR-05-2059. PMID 16489082